CLINICAL TRIAL: NCT01999504
Title: Gut Hormone Response After Two Paleolithic-type Meals Compared to a Modern-type Meal Composed According to WHO Guidelines
Brief Title: Gut Hormone Response After Paleolithic-type Meals
Acronym: FooA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leatherhead Food Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FDS-BNH-1268
Record Dates: First submitted 2013-10-29; First posted 2013-12-03 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Insulin Resistance; Satiety
Keywords: Glucagon-like peptide-1; Glucose-dependent Insulinotropic Peptide; Peptide YY; Glucagon; Satiety; Meal; palaeolithic
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PAL-2 (Experimental): Based on WHO dietary guidelines for protein, fat and carbohydrate but made with ingredients that would have been available in palaeolithic times (e.g. no cereals, no dairy).
  Interventions: Other: PAL-2
- TFH-1 (Experimental): Based on WHO dietary guidelines for protein, fat and carbohydrate but made with ingredients that would have been available in palaeolithic times, (e.g. no cereals, no dairy).
  Interventions: Other: TFH-1
- Reference (Placebo Comparator): Meal based on WHO dietary guidelines for protein, fat and carbohydrate.
  Interventions: Other: Reference

INTERVENTIONS:
Other: PAL-2 — meal
  Arms: PAL-2
Other: TFH-1 — Meal
  Arms: TFH-1
Other: Reference — Meal
  Arms: Reference

SUMMARY:
The effects of two palaeolithic-type meals will be assessed with respect to a panel of gut hormones, satiety, blood glucose and insulin levels as compared to a meal constructed along the lines of the world Health Organisation dietary recommendations

DETAILED DESCRIPTION:
In the current study the effects of two palaeolithic-type meals will be assessed with respect to a panel of gut hormones (including incretins), satiety, blood glucose and insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18-27 inclusive
* Apparently healthy: no medical conditions which might affect study measurements as judged by Leatherhead physician based on a health questionnaire)
* Having general practitioner
* Reported dietary habits: no medically prescribed diet, no slimming diet, used to eat 3 meals a day, no vegetarian
* Reported intense sporting activities less than 10h/w
* Reported alcohol consumption less than 21units/w
* non-smoking
* A fasting capillary blood glucose value within the local normal reference value: 4-6.5 mmol/L measured by finger prick

Exclusion Criteria:

* Use of medication which interferes with the study measurements (as judged by the study physician)
* Being an employee of Unilever or Leatherhead Food Research
* Scoff questionaire score ≥ 2
* Eating habit questionnaire ≥ 14
* Smoking
* Dislike, allergy or intolerance t the test meals or the ad libitum meal
* Reported participation in another nutritional or biomedical trial 3 months before pre-study examination or during the study
* Reported participation in night shift work two weeks prior to the pre-study investigation during the study. Night work is defined as working between midnight and 06.00 AM

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Glucagon-like peptide-1 | 0-3 hours
  Area under the Concentration versus time curve for Glucagon-like peptide-1 in blood plasma

SECONDARY OUTCOMES:
Glucose-dependent Insulinotropic Peptide | 0-3 hours
  Area under the Concentration versus time curve of Glucose-dependent Insulinotropic Peptide in blood plasma
Fullness | 0-4 hours
  Area under the curve for fullness scores (as rated by the subjects on a Visual Analog Scale) versus time
Glucose | 0-3 hours
  Area under the Concentration versus time curve of Glucose in blood
Insulin | 0-3 hours
  Area under the Concentration versus time curve of insulin in blood plasma
Glucagon | 0-3 hours
  Area under the Concentration versus time curve of Glucagon in blood plasma
Peptide YY | 0-3 hours
  Area under the Concentration versus time curve of Peptide YY in blood plasma
Hunger | 0-4 hours
  Area under the curve for hunger scores (as rated by the subjects on a Visual Analog Scale) versus time
Desire to eat | 0-4 hours
  Area under the curve for desire to eat scores (as rated by the subjects on a Visual Analog Scale) versus time

OTHER OUTCOMES:
Insulin/glucose ratio | 30 minutes
  Ratio between insulin and glucose in blood as measured at 30 minutes after start of test product intake
Ad libitum meal | 4 hours
  Weight of an ad libitum pasta with tomato sauce meal consumed at 4 hours after test product intake
Time to return to baseline of satiety score for fullness, hunger and desire to eat | up to 4 hours
  Time to return to baseline for the scores on a Visual Analogue Scales for fullness, hunger and desire to eat
Peptide hormones | 0-3 hours
  Area under the Concentration versus time curve for total amylin, ghrelin, pancreatic polypeptide, C-peptide, leptin, interleukin-6, monocyte chemotactic protein-1 and tumour necrosis factor-alpha in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Diaz-Toledo Trenado, Principal Investigator — Leatherhead Food Research
Locations (1):
- Leatherhead Food Research, Leatherhead, Surrey, United Kingdom